CLINICAL TRIAL: NCT02709421
Title: Risk Factors Related to Post-endoscopic Retrograde Cholangiopancreatography Pancreatitis in High-risk Patients Who Underwent ERCP and Received Prophylactic Rectal Indomethacin
Brief Title: Risk Factors of Post-ERCP Pancreatitis in Patients Receiving Rectal Indomethacin
Status: Completed | Type: Observational
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Yanglin Pan, Associated professor, Air Force Military Medical University, China
Other Study IDs: 20160224-2
Record Dates: First submitted 2016-02-29; First posted 2016-03-16 (Estimated); Last update posted 2016-09-05 (Estimated); Status verified 2016-06

CONDITIONS: Healthy
Keywords: post-Endoscopic Retrograde cholangiopancreatography pancreatitis; Risk factors; Indomethacin

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Indomethacin Group: All the patients with high risks of PEP received administration of one single dose of 100mg rectal indomethacin after ERCP.
  Patients were considered high risk of PEP if they met one of the following criteria: clinical suspicion of sphincter of Oddi dysfunction, a history of PEP, pancreatic sphincterotomy, precut sphincterotomy, ≥8 cannulation attempts, cannulation time≥10 minutes; pneumatic dilatation of an intact biliary sphincter, ≥3 inadvertent pancreatic duct cannulation, opacification of pancreatic acini, or the acquisition of a cytologic specimen from the pancreatic duct with the use of a brush or forceps.

SUMMARY:
Post-endoscopic retrograde cholangiopancreatography(ERCP) pancreatitis (PEP)remains the most frequent adverse event of ERCP. Rectal indomethacin, as one kind of classic NSAIDs, has been proved to be effective in reducing the incidence of PEP. It has been widely used to prevent PEP in patients, especially those with potentially high risks of PEP. However, rectal indomethacin can not completely eradicate the occurrence of PEP. The rate of PEP in patients receiving indomethacin ranges from 3.2% to 9.2%. The risk factors of PEP in patients receiving rectal indomethacin remains unclear. The aim of the study was to identify potential risk factors in high-risk patients whose received administration of prophylactic rectal indomethacin after ERCP.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing diagnostic or interventional ERCP
* Receiving administration of rectal indomethacin(100mg) after ERCP
* High risk patients determined at the discretions of endoscopists

Exclusion Criteria:

* Dose other than 100mg
* Acute pancreatitis within 3 days before ERCP
* Average risk patients at the discretions of endoscopists
* Using NSAIDs within 7 days before ERCP
* Without cannulation attempts
* Administration of rectal indomethacin before or during ERCP

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent ERCP and received administration of rectal indomethacin.
Sampling Method: Non-Probability Sample
Enrollment: 790 (Actual)
Dates: Start 2016-02; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Overall PEP rate | 1 year
  PEP was defined if patients experienced abdominal pain for more than 24h after procedure, accompanying with amylase or lipase ≥ 3 times equal to the upper limit of normal value.

SECONDARY OUTCOMES:
The rate of moderate-severe pancreatitis | 1 year
Overall ERCP-related complication rate | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Yanglin Pan, Principal Investigator — Xijing Hospital of Disgestive Diseases.The Fourth Military University
Locations (3):
- China (3):
  - Department of gastroenterology,Chinese PLA 174 Hospital, Xiamen, Fujian
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Xijing Hospital of Digestive Diseases, Xi'an, Shaanxi

REFERENCES:
- [Background] Dumonceau JM, Andriulli A, Elmunzer BJ, Mariani A, Meister T, Deviere J, Marek T, Baron TH, Hassan C, Testoni PA, Kapral C; European Society of Gastrointestinal Endoscopy. Prophylaxis of post-ERCP pancreatitis: European Society of Gastrointestinal Endoscopy (ESGE) Guideline - updated June 2014. Endoscopy. 2014 Sep;46(9):799-815. doi: 10.1055/s-0034-1377875. Epub 2014 Aug 22. PMID 25148137
- [Background] Yaghoobi M, Rolland S, Waschke KA, McNabb-Baltar J, Martel M, Bijarchi R, Szego P, Barkun AN. Meta-analysis: rectal indomethacin for the prevention of post-ERCP pancreatitis. Aliment Pharmacol Ther. 2013 Nov;38(9):995-1001. doi: 10.1111/apt.12488. Epub 2013 Sep 16. PMID 24099466
- [Derived] Kang X, Zheng L, Zeng W, Yang S, Sun H, Zhang R, Wang X, Wang B, Tao Q, Yao S, Chen J, Pan Y, Guo X. Risk Factors for Post-ERCP Pancreatitis in High-Risk Patients Receiving Post-procedure Rectal Indomethacin. J Gastrointest Surg. 2018 Nov;22(11):1903-1910. doi: 10.1007/s11605-018-3864-0. Epub 2018 Jul 6. PMID 29980976